CLINICAL TRIAL: NCT04339296
Title: Medication Dispensing System to Support Medication Adherence for Individuals Living at Home With Chronic Conditions: A Randomized Controlled Trial
Brief Title: Connected Healthcare for Individuals Living at Home With Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); Catalyst Healthcare Ltd. (Industry)
Responsible Party: Principal Investigator, Mubashir Aslam Arain, Senior Research and Evaluation Consultant, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I2P2-3-00153
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Medication Adherence; Medication Compliance; Medication Nonadherence; Hypertension; Diabetes; Arthritis; Chronic Pain; Anxiety Depression; Asthma
Keywords: Medication dispenser; Medication adherence; Polypharmacy; Chronic conditions; Aging and seniors; Community-dwelling
MeSH Terms: conditions — Medication Adherence; Hypertension; Diabetes Mellitus; Arthritis; Chronic Pain; Asthma; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Participants were assigned to two groups. Intervention participants were assigned to use spencer medication dispenser system. Whereas, control participants continued to use their current method of medication management. Block randomization was used to assign the participants into the intervention or control group as soon as they enrolled in the study. Blocks varied in sizes (10, 12, 14) to reduce the predictability of the allocation assignment within participants and research staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group included medication management with Spencer.
  Interventions: Device: Spencer
- Control Group (No Intervention): The control group continued to use their current method of medication management, such as blister packs, strip packs, pill organizers and plastic prescription vials.

INTERVENTIONS:
Device: Spencer — The MDS dispenses medications on time with visual and audio reminders. The audio alert get louder if the plastic medication packet is not dispensed from the system. The MDS allows participants to dispense their medications early if they are going to be away from home. The system also displays personalized and health-condition speciﬁc questions. The pre-packaged medications are delivered by pharmacy that inserted directly into the spencer device. Spencer system is non-inclusive and approved by Health Canada.
  Other Names: Medication Dispensing System (MDS)
  Arms: Intervention group

SUMMARY:
Managing and taking medications as prescribed can be a difficult task. This is especially true for older adults living at home with chronic conditions while managing multiple prescribed medications. In response, Catalyst Healthcare has adopted an integrated medication dispensing system that intends to improve patient adherence to medications and quality of care through real-time pharmacists and caregiver support.Catalyst Healthcare has launched an integrated at-home medication dispenser system called spencer. Spencer is a natural extension that plugs into Catalyst's AdhereNet platform, connecting high-risk patients in home care setting to a multi-disciplinary care team in real-time. Study is funded by the Centre of Aging and Brain Health Innovation (CABHI).

Investigators are conducting a randomized controlled trial with a target sample size of 100 participants to examine the efficacy of an in-home electronic medication dispensing system (MDS) on improving medication adherence in community-dwelling older adults with chronic conditions. 50 of these participants will be assigned to the intervention group (medication management with Spencer) and 50 will be assigned to the control group (medication management without Spencer). Medication adherence and patient-related data will be collected over a six-month period. Participants health status and characteristics will be obtained through baseline assessment upon enrollment. A monthly follow-up survey will be completed to collect medication management and adherence data. Adherence data for spencer-users will be collected from Catalyst Healthcare technology platform. In the control group, adherence will be measured through monthly medication logs completed by participants.

DETAILED DESCRIPTION:
Purpose: It is estimated by 2045, one in five Albertans in Canada will be 65 or older. Medication compliance in the senior population is a significant challenge for optimizing patient outcomes. This has significant implications when nearly 69% of medication related hospitalizations are attributed to non-adherence and the estimated cost to the Canadian Health care system is $7-$9 billion. The factors that contribute to poor medication adherence are multifactorial. For example, multiple medications within a treatment regimen, increased frequency of medication intake and a prolonged course of drug therapy all contribute to decreased medication adherence. Almost 2/3 of those aged 65 and over take five or more prescription drugs thus increasing the risk of adherence issues.

Therefore, therapeutic management of multiple chronic diseases can only be realized when the individual is adherent to their prescribed pharmacological regimen. Age-related innovations provide an enormous opportunity to enhance the quality of life for seniors and reduce healthcare cost related to medication adherence issues. The spencer medication dispensing device is a new integrated technology that improves medication compliance and offers independence to seniors at home while providing real-time pharmacist and caregiver support. Alberta Health Services (AHS) is committed to supporting and strengthening community care by adopting age-related innovations. Hence, the aim of study is to evaluate user benefits and effectiveness of the device for improving medication compliance in older adults and seniors population.

Primary Research Question: Does the spencer system improve medication adherence in individuals 50 year or older living in the community taking five plus medications?

Study Design: This Randomized Controlled Trial (RCT) with the spencer device will be conducted from March 2019 to June 2020 in Calgary, Alberta. The data will be collected over a six-month period, the spencer deployment will begin in April 2019 and will continue till September 2019. This is a proof of concept study for which no formal sample size calculation is required. A total of 100 study participants will be recruited in the study (50 intervention group and 50 in the control group). The investigators will randomly place a participant in either the intervention group to use spencer or into the control group to continue the using their current method of management.

Randomization: The investigators will be using block randomization which is the recommended method for sample sizes of 50 or less in each group to balance the groups in terms of the number of subjects they contain, and in the distribution of potential confounding variables. The study is not blinded so the blocks will vary in sizes (10, 12, 14) to reduce the predictability of the intervention assignment. A project assistant (a contracted staff which will not be involved in data collection or analysis activities) will produce computer-generated sets of random allocations in advance of the study and then sealed in consecutively numbered opaque envelopes. Once the participants has given consent to be included in the study, he/she will then be irreversibly randomized by opening the next sealed envelope containing his/her assignment.

Technology Intervention: The spencer device comprises interactive tools to optimize medication adherence and clinical outcomes. The device dispenses the patient's medications on time with reminders by sending visual and audio alerts. The sound of the audio alerts get louder if the medication pouch is not removed from the device by the patient. Patient have two hour window to remove the medication pouch. If not removed, patients are considered non-adherent for that particular time frame. Spencer allows individuals to dispense their medication early if away from home. Medication adherence is tracked through spencer Care platform. The medication adherence is based on an assumption that medication was administered by a patient once the pouch was removed from the device.

Also, spencer uses a multi-disciplinary approach of care team members including pharmacists, caregivers and spencer medication adherence platform to provide healthcare in to the homes of the high-risk, chronically-ill population. The device supports a personalized plan that tracks medication adherence and response to therapy. Spencer displays personalized and condition specific questions to meet the individual goals of patients. Patients can respond to disease specific questions in spencer. Spencer certified pharmacists have the ability to review patient responses remotely and determine the need for reassessment, medication reconciliation and clinical intervention as appropriate. Spencer permits intervention remotely through Telehealth capabilities and consultation. Patient receives appointment time directly from spencer, spencer automatically rings at designated time, and call is initiated when patient answers with the touch of a screen. Daily tracking of medication adherence and response to relevant clinical engagement questions will be conducted via the spencer platform.

Through the connected devices, spencer ensures that everyone in the circle of care can participate in the wellbeing of the patient. Spencer Assist is a mobile app that allows caregivers and family members to support patients at home. Medication adherence data is also accessible to the health care team. The pharmacist, health care provider and caregiver are now electronically connected to patients and can access data regarding deviations in adherence in real time. This connectivity allows for earlier intervention to provide the support needed for improved healthcare outcomes.

The spencer system empowers patients to manage their treatment regimen and schedule from the comfort of their own home. Spencer technology addresses key priority areas related to Aging in place, independence, and caregiver support and care coordination with care team and caregivers.

Primary outcome: The study will look at patient focused outcome and seek to understand the influence of the medication dispensing device on medication adherence. Specifically, increased patient medication adherence in the intervention group as a result of spencer utilization. In the intervention group, the medication adherence data will be retrieved from the Catalyst spencer medication adherence platform. In the control group, the medication adherence will be will be self-reported and participants will be required to maintain missed dosage logs. Participants will complete self-reported adherence questionnaire in both groups (intervention and control) at baseline assessment and end of the study for comparison purposes.

Catalyst Healthcare defines Adherence percent as actual pill (s) dispensed from the spencer at the prescribed time within a two hour time window. Average medication adherence will be calculated by an average of all "pill level" adherence numbers i.e. if all pills were taken within the window, the adherence number would only contain 100 values. Alternately if no pills were taken within the window, the adherence number would only contain 0 values. Adherence number for a patient within the time range then divided by the total number of pills will provide average medication adherence. Similar approach will be used for calculating medication adherence for control group participants.

Data source and variables: the investigators will use data from multiple sources: Catalyst technology platform for adherence; determine baseline health status of the participants and characteristics by doing initial assessment upon enrollment; and a monthly follow-up survey will be completed to collect medication management data and record any changes in health status or healthcare needs

Data analysis: Data will be entered and analyzed using Statistical Package for the Social Sciences (SPSS) version 25. Descriptive and inferential statistics will be used to compare the baseline status of the intervention and control group as well as at the end of the intervention period. A Chi-square test of independence will be used for categorical variables such as the number of participants who missed one or more medication dosage in each group. An independent sample t-test will be performed for continuous variables such as to compare the average number of missed medicines between the intervention and control group. Any confounding factors will be controlled in the regression model. Statistical tests for inferential statistics will be set at 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

1. English speakers
2. age 50 and over
3. diagnosed with one or more chronic condition(s) and
4. currently taking ﬁve or more prescribed oral medications.
5. City of Calgary resident

Exclusion Criteria:

* Patients with moderate to severe cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mubashir A Arain, PhD, Principal Investigator — Alberta Health services
Locations (1):
- East Calgary Family Care Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators will be aggregating the data for research purposes and will not release participant-specific data. Also, since this research falls under the auspices of AHS, all data collection, management, and storage processes will fully comply with the Health Information Act and the Freedom of Information and Protection of Privacy Act.

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- [Derived] Arain MA, Ahmad A, Chiu V, Kembel L. Medication adherence support of an in-home electronic medication dispensing system for individuals living with chronic conditions: a pilot randomized controlled trial. BMC Geriatr. 2021 Jan 14;21(1):56. doi: 10.1186/s12877-020-01979-w. PMID 33446126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from a Family Care Clinic during the period of June to October 2019. The clinic mailed invitation letters to potentially eligible participants. Also, potentially eligible participants with scheduled appointments at the clinic were flagged by clinic staff so they could be informed and directed to research staff.
Pre-assignment Details: A total of 91 participants were assessed for eligibility and 50 were randomized into the two groups; 24 allocated to intervention and 26 allocated to control. A total of 16 spencer participants and 17 control participants completed the study. The study dropout rate was 33% (n=8) and 35% (n=9) in the intervention and control group, respectively.
Groups:
- Intervention Group: Intervention group included medication management with Spencer.
  Spencer dispenses medications on time with visual and audio reminders. The audio alert get louder if the plastic medication packet is not dispensed from the system. Spencer allows participants to dispense medications early if they are going to be away from home. The system also displays personalized and health-condition speciﬁc questions. The pre-packaged medications are delivered by pharmacy that inserted directly into the spencer device. Spencer system is non-inclusive and approved by Health Canada.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 24 | 26
Completed Baseline | 23 | 25
Received Allocated Intervention | 21 | 24
Completed | 16 | 17
Not Completed | 8 | 9
Not completed — Refuse to participate after allocation | 1 | 1
Not completed — Withdrew after completion of baseline | 2 | 1
Not completed — Lost to Follow-up | 0 | 4
Not completed — Discontinued intervention | 5 | 3

BASELINE CHARACTERISTICS:
Population: From the 50 participants randomized; 24 were allocated to intervention and other 26 allocated to control. However, one participant in each group refused to participate after allocation and didn't complete the baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.96 (7.86) | 59.92 (5.93) | 61.94 (6.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 21 | 24 | 45
  Aboriginal | 1 | 1 | 2
  South East Asian | 1 | 0 | 1
Living Arrangement [Count of Participants; unit: Participants]
  Alone in residence | 8 | 12 | 20
  With Spouse | 8 | 5 | 13
  With family member(s) other than spouse | 4 | 3 | 7
  Other | 3 | 5 | 8
Education [Count of Participants; unit: Participants] — Population: One intervention participant preferred not to disclose this information.
  Participants
    Less than High School Diploma: number analyzed (Participants) | 22 | 25 | 47
    Less than High School Diploma | 5 | 7 | 12
    High School Diploma: number analyzed (Participants) | 22 | 25 | 47
    High School Diploma | 4 | 6 | 10
    Some College, no degree: number analyzed (Participants) | 22 | 25 | 47
    Some College, no degree | 11 | 7 | 18
    Bachelor's Degree: number analyzed (Participants) | 22 | 25 | 47
    Bachelor's Degree | 2 | 5 | 7
Employment Status [Count of Participants; unit: Participants]
  Employed (Full Time) | 0 | 1 | 1
  Employed (Part Time) | 1 | 0 | 1
  Unemployed | 1 | 2 | 3
  Retired | 11 | 6 | 17
  Disabled | 10 | 16 | 26
Annual Income [Count of Participants; unit: Participants] — Population: One control participant preferred not to disclose this information.
  Participants
    < $21,000: number analyzed (Participants) | 23 | 24 | 47
    < $21,000 | 9 | 16 | 25
    $21,000 - $40,000: number analyzed (Participants) | 23 | 24 | 47
    $21,000 - $40,000 | 9 | 6 | 15
    > $41,000: number analyzed (Participants) | 23 | 24 | 47
    > $41,000 | 5 | 2 | 7
Chronic Health Conditions [Mean (Standard Deviation); unit: Chonic conditions] | 4.48 (2.19) | 4.20 (1.98) | 4.34 (2.09)
Prescribed Medications [Mean (Standard Deviation); unit: Prescribed medications] | 9.39 (3.73) | 10.12 (4.76) | 9.76 (4.25)
Over-the-counter (OTC) Medications [Mean (Standard Deviation); unit: OTC medications] | 1.68 (1.84) | 2.12 (2.74) | 1.90 (2.29)
Help Taking Medication [Count of Participants; unit: Participants] — Question - Do you require any form of help with taking your medications (i.e., reminder, physical assistance, organizing or sorting medication…etc)?
  Participants
    Yes | 5 | 4 | 9
    No | 18 | 21 | 39
Medication Management Method [Count of Participants; unit: Participants] — Question - What is your current method of medication management? Population: Some participants in both groups didn't know about their medication management method and response wasn't recorded.
  Participants
    Blister Pack: number analyzed (Participants) | 19 | 23 | 42
    Blister Pack | 5 | 12 | 17
    Pill Organizers: number analyzed (Participants) | 19 | 23 | 42
    Pill Organizers | 9 | 4 | 13
    None (pill containers): number analyzed (Participants) | 19 | 23 | 42
    None (pill containers) | 2 | 6 | 8
    Other: number analyzed (Participants) | 19 | 23 | 42
    Other | 3 | 1 | 4
Medication Times/Day [Mean (Standard Deviation); unit: Number of medication times per day] — Question - How many times a day do you take your prescribed medications?
  Number of medication times per day | 2.91 (0.92) | 2.87 (1.11) | 2.89 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Recorded Medication Adherence
Description: The intervention group adherence recording was obtained from Catalyst's AdhereNet platform. The spencer adherence was defined as percentage of medications dispensed from the system at the prescribed time. The user had a two-hour window to remove the medication pouch. If dispensed, they are given a score of 100 for the particular medication time. If not removed, the user was considered non-adherent and given a score of 0. Weekly medication adherence was calculated by taking the seven day average of daily dispensing adherence values. In the control group, adherence was measured through monthly medication calendars completed by participants. Each participant received customized calendars based on their medications timings along with instruction sheet for tracking their medications. Participants were required to mark "X" on the calendar on the day and time they missed taking their medication(s). Average adherence (weekly) was used as a primary outcome measure.
Time Frame: 26 weeks
Population: Intention-to-treat analysis was utilized. From the 21 intervention participants that started using spencer, adherence data was only collected from 20 participants. One participants withdrew right after receiving spencer and no data was collected. From 24 control participants, no adherence data was collected from two lost to follow participants.
Measure: Mean (Standard Deviation); unit: percentage of medication adherence
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 22
percentage of medication adherence | 98.35 (2.15) | 91.17 (9.76)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Equivalence — An independent sample t-test was performed between intervention and control group to determine if the difference of the mean medication adherence is equal to zero (null hypothesis); p < 0.01, t-test, 2 sided — Statistical test was set at 95% confidence level; Mean Difference (Net) = 7.18 — Medication Adherence Difference = Intervention Adherence - Control Adherence

2. Primary Outcome: Self-reported Medication Adherence
Description: The within group difference in mean rating scores of self-reported medication adherence. The adherence question asked participants to rate their medication adherence on a scale of 1 (non-adherent) to 10 (adherent).
Time Frame: 6-months
Population: Paired sample t-test completed was used at baseline (pretest) and six-month (posttest) for intervention and control group. In the intervention group, adherence data was collected from 16 participants who completed the study. In the control group, 17 participants completed the study but six-month data wasn't collected from two participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 15
score on a scale
  Baseline (Pretest) | 7.63 (1.63) | 7.20 (1.74)
  6-month (Posttest) | 9.13 (0.81) | 8.27 (2.09)
Statistical Analysis 1: Comparison: Intervention Group; Test type: Equivalence — The null hypothesis assumes that the true mean difference for intervention participants self-reported medication adherence scores (from baseline to 6-month) is equal to zero; p < 0.01, t-test, 2 sided — Statistical test was set at 95% confidence level; Mean Difference (Net) = -1.50 — Mean difference (intervention participants self-reported score) = baseline minus 6-month
Statistical Analysis 2: Comparison: Control Group; Test type: Equivalence — The null hypothesis assumes that the true mean difference for control participants self-reported medication adherence scores (from baseline to 6-month) is equal to zero; p = 0.07, t-test, 2 sided — Statistical tests was set at 95% confidence level; Mean Difference (Net) = -1.07 — Mean difference (control participants self-reported score) = baseline minus 6-month

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Intermittent data collected because some participants were unavailable for all monthly follow-up phone calls; control participants were not consistently sending in tracking calendars; intervention participants experienced some technical issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04339296/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04339296/SAP_002.pdf
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT04339296/ICF_003.pdf